CLINICAL TRIAL: NCT02103010
Title: Predictive Modelling for Patient Stratification According to Treatment-related Toxicity and Survival After Chemoradiation for Head and Neck Cancer
Acronym: PRETOXIS
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other); Universitaire Ziekenhuizen KU Leuven (Other); Maastro Clinic, The Netherlands (Other); Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/895
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HNC patients: head and neck cancer patients

SUMMARY:
Radiotherapy is an integral component of the current multimodality treatment approach in locally advanced head and neck cancer (HNC). There is growing evidence that more aggressive treatment regimens improve tumour control and survival. However, intensified treatment is at the expense of increased toxicity, in particular severe acute mucositis. In addition and of increasing importance, late and irreversible treatment-related side effects, including xerostomia and swallowing dysfunction, occur in a considerable proportion of patients and negatively affect quality of life.

High-risk human papilloma virus (HPV), specifically HPV type-16, is implicated as the causative factor in a proportion of HNC, especially those of the oropharynx. HPV-related cancers respond well to chemoradiotherapy compared to HNC related to tobacco and alcohol. Furthermore, the incidence of HPV-related oropharyngeal cancer is rising in Western countries. Given the significant toxicity associated with concurrent chemoradiotherapy, subsets of patients could be managed differently.

The first objective of the project is to develop predictive models for radiation-induced dysphagia and xerostomia in HNC patients. Clinical characteristics, treatment parameters, dose-volume effects on healthy tissues and whole-genome genetic data will be considered. The second objective of the project is to study the prognostic value of HPV status together with a panel of tumour biomarkers in oropharyngeal cancer patients. The overall aim of the project is to stratify patients according to the risks (side-effects) and benefits (survival) of cancer treatment using the developed risk models. Clustering patients into different risk categories may aid treatment decision making reducing therapy toxicity without compromising survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of oral cavity, oropharynx, hypopharynx and larynx. Histologically confirmed cervical lymph node metastases of unknown primary cancer (CUP). For prognosis part of the study: only histologically confirmed squamous cell carcinoma of the oropharynx

  * Stages : Tany N1-3, T3-4 N0, T1-2 N0, if prophylactic neck irradiation is performed
  * Multidisciplinary decision of curative radiotherapy or radiochemotherapy
  * Karnofsky performance status ≥ 70%
  * Age ≥ 18 years old
  * Gender : male - female
  * Informed consent obtained, signed and dated before start of radiotherapy

Exclusion Criteria:

* Treatment combined with brachytherapy
* Treatment combined with cetuximab or other targeted agents
* Prior irradiation to the head and neck region
* History of prior malignancies, except for cured non-melanoma skin cancer, curatively treated in-situ carcinoma of the cervix or other cancer curatively treated and with no evidence of disease at least 5 years
* Distant metastases
* Pregnant or lactating women
* Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study
* Patients unlikely to comply with the protocol, i.e. uncooperative attitude, inability to return for follow-up visits, and unlikely to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with head and neck cancer
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in dysphagia | during radiotherapy and at 6/12/18/24 months after the end of radiotherapy
  Dysphagia during radiotherapy and at 6/12/18/24 months after the end of radiotherapy using the CTCAE (Common Terminology Criteria for Adverse Events) v4.0 scale.
change in xerostomia | during radiotherapy and at 6/12/18/24 months after the end of radiotherapy
  xerostomia during radiotherapy and at 6/12/18/24 months after the end of radiotherapy using the CTCAE (Common Terminology Criteria for Adverse Events) v4.0 scale
change in overall survival | up to three years after study start
change in disease specific survival | up to three years after study start
change in progression-free survival | up to three years after study start
appearance of distant metastasis | up to three years after study start

SECONDARY OUTCOMES:
Change in weight loss | during radiotherapy and at 6/12/18/24 months after the end of radiotherapy
change of Quality of life | pre-radiotherapy, at the last day of radiotherapy and post-radiotherapy (12/24 months)
  using the EORTC (European Organisation for Research and Treatment of Cancer ) quality of life questionnaire C30 and the hand and neck cancer specific quality of life questionnaire HN35

CONTACTS AND LOCATIONS:
Overall Officials: Kim De Ruyck, Dr., Principal Investigator — Ghent University - Department of Basic Medical Sciences
Locations (2):
- Belgium (2):
  - Department of Radiotherapy, University Hospital Ghent, Ghent
  - Department of Radiotherapy, University Hospital Leuven, Leuven